CLINICAL TRIAL: NCT06351761
Title: Validation of Withings BeamO With Withings ECG-App for the Detection of Atrial Fibrillation
Brief Title: WIBOFA - Validation of SCT02 With ECG-App for Detection of AF
Acronym: WIBOFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SCT02-ECG
Record Dates: First submitted 2024-03-13; First posted 2024-04-08 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Normal Sinus Rhythm (Experimental): Simultaneous ECG recording of patient with Normal Sinus Rhythm with investigational and reference devices
  Interventions: Device: Investigational Device (Withings SCT02) 30 second Electrocardiogram recording; Device: Reference Device (Schiller Cardiovit FT-1) 30 second Electrocardiogram recording
- Atrial Fibrillation (Experimental): Simultaneous ECG recording of patient with Atrial Fibrillation with investigational and reference devices
  Interventions: Device: Investigational Device (Withings SCT02) 30 second Electrocardiogram recording; Device: Reference Device (Schiller Cardiovit FT-1) 30 second Electrocardiogram recording
- Arrhythmia other than Atrial Fibrillation (Experimental): Simultaneous ECG recording of patient with Arrhythmia other than Atrial Fibrillation with investigational and reference devices
  Interventions: Device: Investigational Device (Withings SCT02) 30 second Electrocardiogram recording; Device: Reference Device (Schiller Cardiovit FT-1) 30 second Electrocardiogram recording

INTERVENTIONS:
Device: Investigational Device (Withings SCT02) 30 second Electrocardiogram recording — 30 second ECG recording with investigational device (Withings SCT02)
Device: Reference Device (Schiller Cardiovit FT-1) 30 second Electrocardiogram recording — 30 second ECG recording with reference device (Schiller Cardiovit FT-1)

SUMMARY:
The aim of the study is to evaluate the performance of Withings SCT02 with embedded Withings ECG-app in the automatic detection of atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Male or female who are 22 years of age or older
* Subject able to read, understand, and provide written informed consent
* Subject willing and able to participate in the study procedures as described in the consent form
* Subject able to communicate effectively with and willing to follow instructions from the study staff

Exclusion Criteria:

* Subject with an implanted electrical device (i.e. pacemaker, ICD …), whether active or inactive
* Pathologic disorders that may affect motricity resulting in significant hands tremor that prevents subject from being able to hold still (e.g. Parkinson disease)
* Myocardial Infarction (MI) within 90 days prior to the enrollment
* Pulmonary embolism or pulmonary infarction within 90 days prior to the enrollment
* Stroke or Transient Ischemic Attack (TIA) within 90 days prior to the enrollment
* Active or history of life-threatening rhythms as determined by investigators (e.g. ventricular tachycardia, ventricular fibrillation, 3rd degree heart block)
* Any cardiovascular disease that investigators would consider as a risk to subject or renders data uninterpretable (e.g. recent or ongoing unstable angina, decompensated heart failure, active myocarditis or pericarditis)
* Active or symptomatic skin disease on Schiller electrode attachment sites or fingertips which would be in contact with BeamO electrodes (e.g. eczema, rosacea, impetigo, dermatomyositis or allergic contact dermatitis)
* Known sensitivity to medical adhesives, isopropyl alcohol,, electrocardiogram (ECG) electrodes, including known allergy or sensitivity to stainless steel (used in BeamO electrodes).

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 371 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Co-primary outcome 1 - Sensitivity of Investigational Device | 10 months
  Sensitivity (percentage of true positives) in detecting AF from conclusive recordings generated by the software under test, that is recordings resulting in a classification of AF or SR by the IMD, compared to the reference 12-lead ECG.
Co-primary outcome 2 - Specificity of Investigational Device | 10 months
  Specificity (percentage of true negatives) in detecting AF from conclusive recordings generated by the software under test, that is recordings resulting in a classification of AF or SR by the IMD, compared to the reference 12-lead ECG.

SECONDARY OUTCOMES:
Rhythm classification by ranges of heart rate | 10 months
  On pairs of strips such that the rhythm classification of the 12-lead ECG is either SR or AF and such that the strip generated by the IMD is classified as either SR or AF, the classification into four heart rate subgroups will be evaluated.
  * Sinus Rhythm, (50-99 bpm)
  * High Heart Rate (No signs of AFib) (100-150 bpm)
  * Atrial Fibrillation (50-99 bpm),
  * Atrial Fibrillation (100-150 bpm)
Quality of plots measured by the IMD - ECG Waveform Visibility | 10 months
  Clinical Equivalence of ECG waveforms will be qualitatively and quantitatively assessed between the 1-lead generated by the IMD and the lead I of the 12-lead reference ECG determined by certified cardiologists. Equivalence will be evaluated by FV : Fraction of concordant assessments of visibility between the IMD and the reference
Quality of plots measured by the IMD - ECG Waveforms Polarity | 10 months
  On waveforms with waves that are Visible, Clinical Equivalence of ECG waveforms will be qualitatively and quantitatively assessed between the 1-lead generated by the IMD and the lead I of the 12-lead reference ECG determined by certified cardiologists. Equivalence will be evaluated by FP : Fraction of concordant assessment of polarity between IMD and reference
Quality of plots measured by the IMD - ECG Waveforms Intervals | 10 months
  Determine the equivalence of PR, QRS and QT intervals durations between the lead I of the IMD and the lead I of the reference ECG determined by an independent board of certified cardiologists. Duration error will be calculated.
Quality of plots measured by the IMD - Heart Rate calculation | 10 months
  Determine the equivalence of the heart rate (HR) calculated by the IMD and the HR measured by an independent board of certified cardiologists or cardiology technicians on the ECG of the reference.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - FWD Clinical Research, Boca Raton, Florida
  - Diverse Clinical Research, Miami, Florida
- France (2):
  - Henri Mondor University Hospital, Créteil, Val De Marne
  - Centre Cardiopole Trubert, Paris

IPD SHARING:
Plan to Share IPD: No